CLINICAL TRIAL: NCT02686775
Title: The PACO Project: A Randomized Clinical Study of a PAtient COach Program in Vulnerable Lung Cancer Patients
Brief Title: The PACO Project: A Clinical Study of a PAtient COach Program in Vulnerable Lung Cancer Patients
Acronym: PACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Cancer Society (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Oksbjerg Dalton, Senior Researcher, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R73-A4769-13-S17
Record Dates: First submitted 2016-01-21; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer; Social Inequality
MeSH Terms: conditions — Lung Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient coach (Experimental): Standard care and patient coach. 5 face-to-face sessions of approximately 1-2 hours duration and 3 phone calls from inclusion to one month after end of first line treatment. Deviations from this schedule might depend on the treatment modules and on the wishes and needs of the patient. Several patients will continue directly into palliative care and the coach will thus support this transition.
  Interventions: Behavioral: Patient coach; Behavioral: Standard care
- Standard treatment (Active Comparator): Standard care.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Patient coach
  Arms: Patient coach
Behavioral: Standard care

SUMMARY:
The randomized trial evaluates whether assigning a patient coach to vulnerable lung cancer patients will empower these patients to participate in the treatment decision process, help patients navigate the health care system while undergoing treatment and adhere to cancer treatment and to recommendations for supportive care. Half of the participants will receive standard care and be offered a patient coach while the other half will receive standard care.

DETAILED DESCRIPTION:
Having short education or living without a partner negatively influences lung cancer survival and low social position has been associated with higher risk of advanced stage of the lung cancer at diagnosis. Disparities exists in both curative and palliative intended treatment, even adjusted for performance status and comorbidity. Differences in stage, treatment and comorbidity at diagnosis explain most of the social inequality in lung cancer survival. Age disparities in favor of younger lung cancer patients has also been found in several studies showing that older patients do not receive the most optimal treatment although age by itself do not worsen efficacy or tolerance to combined induction and definitive treatment, radiation therapy or concurrent chemoradiation. Taken together these findings indicate that in order to reduce social inequality in lung cancer survival not only early detection should be improved but also efforts to ensure optimal treatment among lung cancer patients of low social position are needed. Survival observed in the most advantaged group of lung cancer patients should set the target for what is achievable for all lung cancer patients in Denmark.

In the present intervention the investigators bring navigation together with activation as a longitudinal intervention by assigning a patient coach to vulnerable lung cancer patients while undergoing treatment. The patient coach function will address patient barrier factors, provider factors and organizational factors through providing social support, practical assistance and linking with health personnel, which are the three main principles guiding the coach intervention. The intervention will target specific phases in the treatment trajectory, which include challenges to compliance: into treatment, maintaining treatment and finalizing treatment. The investigators will use patient coaches who are volunteers with health education to provide a support function that is affiliated to the patient. The investigators believe that assistance with navigating the system, communication with health staff and social support across care transitions will help patients to obtain best possible care Primary aim: optimal treatment depending on stage, histology and performance status Secondary aims: quality of life and symptoms, participation in self-management plans as smoking cessation, physical activity, dietary changes, and short-term survival.

The investigators expect that compared to the usual care group the intervention group will initiate and adhere more to optimal treatment according to stage and performance status. Further, compared to the usual care group the intervention group will report better quality of life, less symptoms related to disease and treatment, higher level of adherence to recommendations for smoking, diet and exercise and better survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-small cell lung cancer or small cell lung cancer
* Referred for further treatment at the oncology ward OR
* Must either 1) Live alone (irrespective of education) or 2) Have no formal education beyond secondary school, or 3) Have one or more comorbidities, or 4) a performance status of 1-2, or 5) be more than 65 years old at time of inclusion.

Exclusion Criteria:

* Dementia
* Being institutionalized
* No proficiency of Danish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Receipt of first-line treatment according to clinical guidelines reported as a binary variable (yes/no) | 20 weeks
  Optimal first line treatment will be defined according to TNM status and performance status and categorized receipt of first-line treatment as binary variable (yes/no).

SECONDARY OUTCOMES:
Differences between groups in overall quality of life using the generic EORTC QLQ-C30 questionnaire (overall quality of life and functioning levels) and the lung cancer specific questionnaire QLQ-LC13 (symptoms) | Then questionnaire will be distributed 3 times: 1) At treatment start (inclusion and baseline assessment), 2) end of treatment, approx. 20- 24 weeks after start of treatment (FU1) 3) one month after end of first line treatment (FU2)
Differences between groups in patient knowledge, skill, and confidence for self-management as assessed by the Patient Activation Measure (PAM) questionnaire | The questionnaire will be distributed 3 times: At treatment start (inclusion and baseline assessment), 2) end of treatment, approx. 20- 24 weeks after start of treatment (FU1) 3) one month after end of first line treatment (FU2)
Differences between groups in patients beliefs in the ability to deal efficiently with a wide range of stressors as assessed by the General Self-Efficacy Scale questionnaire | The questionnaire will be distributed 3 times: At treatment start (inclusion and baseline assessment), 2) end of treatment, approx. 20- 24 weeks after start of treatment (FU1) 3) one month after end of first line treatment (FU2)
Participation in self-management plans regarding smoking cessation reported as binary variable (yes/no) as assessed by a study specific questionnaire and medical records | The outcome will be assessed at FU2 (one month after end of first line treatment)
Differences between groups in depression and anxiety as assessed by the Hospital Anxiety and Depression Scale (HADS) | The questionnaire will be distributed 3 times: At treatment start (inclusion and baseline assessment), 2) end of treatment, approx. 20- 24 weeks after start of treatment (FU1) 3) one month after end of first line treatment (FU2)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne O Dalton, Senior researcher, Principal Investigator — Danish Cancer Society Research Center
Locations (1):
- Department of Oncology, Herlev Hospital, Herlev, Herlev, Denmark